CLINICAL TRIAL: NCT04714632
Title: Vestibular Function in Adolescents With Idiopathic Scoliosis
Brief Title: Function of Inner Ear Such as Balance and Perception of Verticality in Children With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Klara Kucerova, Master of science, Charles University, Czech Republic
Other Study IDs: 260119
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Idiopathic Scoliosis; Vestibular Abnormality
Keywords: idiopathic scoliosis; subjective visual vertical; vestibular evoked myogenic potentials; posturography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with idiopathic scoliosis: Adolescent between 10-18y with diagnosing idiopathic scoliosis
- Healthy children: Healthy children between 10-18y without any orthopedics problems

SUMMARY:
The purpose of this study was to evaluate vestibular function in children with idiopathic scoliosis as a possible cause of etiopathogenesis of its diagnose.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic scoliosis

Exclusion Criteria:

* operation of the spine
* neurological disease
* hearing problems

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with Idiopathic scoliosis
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Vestibular evoked myogenic potentials | up to 6 months
  To evaluate the results of vestibular evoked myogenic potentials we used the latency (ms) and the amplitude (μV) of the positive wave (P13) and the negative wave (N23)
Posturography | up to 6 months
  Posturography was measured in 6 different sensory conditions. The posturographic parameters of center of pressure were measured for this study.
Perception of subjective visual vertical | up to 6 months
  We measured perception of subjective visual vertical (SVV) in static and dynamic conditions. Each participant completed a total of six trials for static SVV and twelve trials for dynamic SVV, in six trials the optokinetic background rotated clockwise and in six trials counterclockwise. Norms for static conditions are ±2° and for dynamic conditions ±4°

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation and Sports Medicine, University Hospital Motol, Prague, Czechia